CLINICAL TRIAL: NCT01181245
Title: A Phase 1 Study of Safety and Bioactivity With FG-3019 in Combination With Gemcitabine and Erlotinib for Subjects With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-MC3019-028
Record Dates: First submitted 2009-05-04; First posted 2010-08-13 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Locally Advanced or Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pamrevlumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FG-3019 (Experimental): All subjects are treated with FG-3019
  Interventions: Drug: FG-3019

INTERVENTIONS:
Drug: FG-3019 — 3mg/kg IV, 10mg/kg IV, 15mg/kg IV, 25mg/kg, 35mg/kg IV, 45mg/kg IV - Biweekly, 35/17.5mg/kg, 45/22.5 mg/kg - Weekly

SUMMARY:
Objectives

* Primary: To evaluate the safety and tolerability of FG-3019 in combination with gemcitabine and erlotinib
* Secondary: To evaluate the efficacy and pharmacokinetics of FG-3019 in combination with gemcitabine and erlotinib

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent
2. Males and females aged ≥18 years old
3. Histologically or cytologically confirmed adenocarcinoma of the pancreas
4. Locally advanced (Stage III) or metastatic (Stage IV) adenocarcinoma of the pancreas
5. Spiral CT scan demonstrating at least one pancreatic adenocarcinoma measurable lesion according to RECIST criteria and PET scan showing metabolically active lesion (for the last six subjects in the 15 mg/kg and the subjects in the 25 mg/kg FG-3019 dose cohorts only)
6. Women of childbearing potential and men must use effective contraception during and for at least 90 days following study participation. Women of childbearing potential must have a negative Screening serum pregnancy test.
7. ECOG performance status score of 0-1
8. Life expectancy >12 weeks
9. Ability to adhere to the study visit schedule and understand and comply with all protocol requirements and instructions from study staff

Exclusion Criteria

1. Absolute neutrophil count (ANC) <500 cells/mm3
2. Hemoglobin <10.0 g/dL
3. Platelet count <100,000 cells/mm3
4. Bilirubin >2.0 x upper limit of normal (ULN)
5. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2.5 x ULN, or >3.5 x ULN if liver metastases are present
6. If the subject is diabetic, HbA1c >10%
7. Current pregnancy or breast feeding due to recent pregnancy
8. History of another malignancy in the past 2 years with the exception of basal cell or squamous cell carcinoma of the skin
9. Previous chemotherapy with gemcitabine
10. Previous systemic antineoplastic agent (other than adjuvant 5-fluorouracil as radio-sensitizer)
11. Adjuvant 5-fluorouracil within 28 days prior to Day 1
12. Major surgery within 28 days prior to Day 1 (stent placement is allowed)
13. Radiation therapy within 28 days prior to Day 1
14. Clinical evidence or any history of brain metastasis
15. Uncontrolled hypertension (systolic blood pressure [SBP] >180 mmHg or diastolic blood pressure [DBP] >105 mmHg)
16. New York Heart Association Class III or IV congestive heart failure
17. History of allergic or anaphylactic reaction to human, humanized, or chimeric monoclonal antibodies
18. Current clinical or laboratory evidence of active infection requiring antibiotic or antiviral therapy
19. Active major gastrointestinal bleeding
20. Full-dose heparin therapy within 28 days prior to Day 1
21. Participation in studies of investigational products within 42 days prior to Day 1
22. Clinically significant and uncontrolled medical condition considered a high risk for participation in an investigational study or a likelihood that the subject will be unable to comply with protocol requirements and complete the trial (e.g., emphysema requiring supplemental oxygen, poorly controlled arrhythmia, psychiatric illness, Alzheimer's disease)
23. Current abuse of alcohol or drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of FG-3019 in combination with gemcitabine and erlotinib | Through the end of the study

SECONDARY OUTCOMES:
FG-3019 PK parameters | Through the end of the study
Time to Progression (TTP) | Through the end of the study
6-month, 12-month and overall median survival rates | Through the end of the study
Maximal tumor response as determined by RECIST criteria | Through the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Albert C Koong, MD, PhD, Principal Investigator — Stanford University; J. Marc Pipas, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Vincent J Picozzi, MD, PhD, Principal Investigator — Virginia Mason Hospital/Medical Center; Peter J O'Dwyer, MD, Principal Investigator — University of Pennsylvania; Smitha Krishnamurthi, MD, Principal Investigator — University Hospitals of Cleveland, Case Comprehensive Cancer Center; Charles Lopez, MD, Principal Investigator — Oregon Health and Science University; Nathan Bahary, MD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - Stanford University School of Medicine, Stanford, California
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University Hospitals of Cleveland, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Oregon Health Sciences University (OHSU), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington